CLINICAL TRIAL: NCT04022421
Title: The Efficacy of Hydroxychloroquine on Behcet's Disease Thrombotic Events Prevention
Brief Title: Hydroxychloroquine Efficacy on Behcet's Disease Thrombosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Abdelkhalik Ahmed Mohamed, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 17300279
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Behcet's Syndrome, Vascular Type
MeSH Terms: conditions — Behcet Syndrome | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- hydroxychloroquine arm (Experimental)
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine — the drug will be taken by one group of the patients daily at a dose of 400mg

SUMMARY:
Patients diagnosed with Behcet's disease will be randomized to administeration of hydroxychloroquine. Assessment will be done for the patients at baseline and every one month in the first three months and then quarterly for one year.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with Behcet's disease on any DMARDs

Exclusion Criteria:

* Patients with critical conditions
* Patients with hypersensitivity or adverse drug reactions to hydroxychloroquine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Prevention of the recurrence of thrombotic events | 6 months- one year
  number of relapses is expected to fall with the longterm use of the drug

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt